CLINICAL TRIAL: NCT07061054
Title: Safety and Efficacy of the CE-Marked NetrodTM Renal Denervation System in Treating Patients With Primary Hypertension in the Absence of Anti-hypertensive Medication: a Pilot Study With 20 Subjects
Brief Title: Netrod-Pilot Study of Renal Denervation With NetrodTM Sixelectrode Radiofrequency RDN System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Golden Leaf MedTec Co. Ltd (Industry)
Collaborators: North American Science Associates Ltd. (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Netrod OFF-MED Pilot
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Uncontrolled Hypertension
Keywords: Renal denervation (RDN); Radiofrequency renal denervation; Sympathetic nervous system; Interventional therapy; Interventional cardiology; Device-based therapy; Renal artery denervation; Blood pressure; Resistant Hypertension; Refractory Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renal Denervation (Experimental): Renal angiogram and Renal Denervation procedure
  Interventions: Device: Netrod™ six-electrode radiofrequency renal denervation system

INTERVENTIONS:
Device: Netrod™ six-electrode radiofrequency renal denervation system — Netrod™ renal denervation (RDN) system, which is indicated for the treatment of uncontrolled hypertension. It consists of the following two components: Netrod™ Six-Electrode Basket Radiofrequency Renal Denervation Catheter and Netrod™ Renal Denervation Radiofrequency Generator. The catheter's electrodes deploy into a self adaptive basket structure, optimizing contact with the vessel wall for effective ablation.

SUMMARY:
This single-arm, non-randomized, open-label investigation aims to collect safety and efficacy data of the CE-Marked Netrod™ RDN System in treating European patients with primary hypertension in the absence of anti-hypertensive medication.

DETAILED DESCRIPTION:
This is a prospective, single-arm, non-randomized, open-label, multi-center study to collect safety and efficacy data of the CE-Marked Netrod™ RDN System in treating European patients with primary hypertension in the absence of anti-hypertensive medication. This clinical investigation aims to enroll 20 patients in Europe. Patients with uncontrolled primary hypertension (office BP ≥150/90 mmHg and <180/110 mmHg) who are willing to discontinue antihypertensive medications will be screened after providing informed consent.

All eligible patients will undergo a medication washout period of at least 21 days, and those who continue to meet the eligibility requirements will undergo the RDN procedure using the Netrod™ RDN System. Subjects will be evaluated at hospital discharge and at 1, 3, 6, and 12 months post-procedure. All subjects will remain off antihypertensive medications until the primary endpoint is assessed at the 3-month follow-up visit, after which antihypertensive medications may be reintroduced.

The primary efficacy endpoint is the change in daytime ambulatory systolic blood pressure (ASBP) from baseline at three months post-procedure. The primary safety endpoint is the incidence of periprocedural major adverse event (MAE) rate through 30 days post index procedure.

ELIGIBILITY:
Inclusion criteria:

1. Subject with age ≥18 years or minimum age as required by local regulations and ≤ 70 years old at time of consent
2. Subject with hypertension who has an office BP of ≥ 150/90 mmHg and < 180/110 mmHg (meet both SBP and DBP criteria) at Screening V2, and mean daytime ASBP ≥ 140 mmHg and < 170 mmHg by 24-hour ABPM at Screening V2.
3. Willing and able to provide informed consent
4. Willing and able to comply with all study-specific visits, assessments, and requirements

Exclusion Criteria:

1. 1. Subject who is pregnant, nursing or planning to become pregnant during the course of the study
2. Subject with unilateral or bilateral renal artery that are not suitable for ablation procedure (renal artery stenosis more than 50%, renal aneurysm, renal artery abnormality, renal artery diameter < 3 mm or treatable segment length < 20 mm)
3. Subject with single-kidney or history of kidney transplant
4. Subject with history of renal artery intervention (Percutaneous Transluminal Angioplasty [PTA] or stenting) or Renal Denervation (RDN)
5. Subject with any conditions that may affect the accuracy of blood pressure (BP) measurement: such as the diameter of the upper arm is too large for the cuff, or arrhythmia, etc
6. Subject with known secondary hypertension
7. Subject with eGFR <40 mL/min/l.73m²
8. Subject with history of hospitalization for hypertensive emergency within past year
9. Subject with type I diabetes mellitus
10. Subject with primary pulmonary hypertension
11. Subject with history of bleeding diathesis and haematological disorders or coagulopathy
12. Subject with recent history of any embolism within 6 months
13. Subject with history of coronary artery intervention, unstable angina or myocardial infarction
14. Subject with stable angina and therefore treated anti-anginal medication (betablockers, calcium antagonists, long-acting nitrates)
15. Subject with history of abdominal aortic aneurysm
16. Subject with atrial fibrillation or history of atrial fibrillation in the last 3 years or on rate or rhythm control medication for arrhythmia
17. Subject with a history of ventricular fibrillation or ventricular tachycardia
18. Subject known with serum Human Immunodeficiency Virus (HIV)-positive
19. Subject who is allergic to contrast agents and not responding to preventive medication
20. Subject with acute or severe systemic infections
21. Subject with mental illness or any psychological problems that may interfere with participating in the study
22. Subject with history of stroke or transient ischemic attack (TIA)
23. Subject with malignant tumors or end-stage disease
24. Subject with severe Peripheral Artery Disease (PAD) along the access path to renal arteries, including abdominal aneurysm
25. Subject with severe heart valve stenosis or regurgitation
26. Subject with heart failure requiring medications (i.e. Angiotensin-Converting Enzyme (ACE)/ Angiotensin II Receptor Blockers (ARB), Sodium-Glucose Cotransporter 2 Inhibitors (SGTL2i), diuretics)
27. Subject with uncontrolled hyperthyroidism or hypothyroidism
28. Subject with severe electrolyte abnormalities, defined as values above and below the limits of normal (LN) on repeated measurements despite normalization efforts, or with liver function abnormalities, defined as 2 > Upper Limit of Normal (ULN)
29. Subject who requires mechanical ventilation other than Continuous Positive Airway Pressure (CPAP) for sleep apnea
30. Subject with an implanted pacemaker or Implantable Cardioverter Defibrillator (ICD)/ Cardiac Resynchronization Therapy (CRT) device
31. Subject with a history of major surgery or trauma within 30 days prior to enrolment
32. Subject who has planned surgery or cardiovascular intervention within the next 12 months
33. Subject who is participating in other drug or medical device clinical investigations
34. Subject who is unsuitable to participate in this study in the opinion of investigators (e.g., drug use or alcohol dependency, cognitive impairment, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of periprocedure major adverse event (MAE) | Through 30 days post index procedure
  Incidence of periprocedure major adverse event (MAE), defined as a composite of the following events through 30 days post index procedure (except for new renal artery stenosis):
  * All-cause mortality
  * End-stage renal disease (ESRD) defined as stage 5 Chronic Kidney Disease (CKD) (Estimated Glomerular Filtration Rate (eGFR) < 15 mL/min/l.73m²) or hemodialysis
  * Significant embolic event resulting in end-organ damage
  * Renal artery perforation or dissection requiring intervention
  * Major vascular complications requiring medical or surgical intervention
  * Hospitalization for hypertensive crisis (unless clearly demonstrated to be associated with non-adherence with antihypertensive medications in the subjects on escape medication)
  * New renal artery stenosis > 70% (must be confirmed by angiography)
Mean daytime ambulatory systolic blood pressure (ASBP) | From baseline to 3 months post index procedure
  Changes from baseline in mean daytime ambulatory systolic blood pressure (ASBP) by 24-hour ambulatory blood pressure monitoring (ABPM) at 3 months post index procedure

SECONDARY OUTCOMES:
Incidence of the safety events | At 3, 6 and 12 months post procedure
  Incidence of the following events:
  * All-cause mortality
  * ESRD defined as stage 5 CKD (eGFR < 15 mL/min/l.73m²)
  * ≥50% decline in eGFR or >50% increase in serum creatinine from baseline
  * New myocardial infarction or acute coronary syndrome (ACS)
  * New stroke or Cerebrovascular Accident (CVA)
  * Renal artery reintervention
  * New renal artery stenosis > 70% confirmed by angiography
  * Hospitalization for hypertensive crisis not related to confirmed non-adherence of anti-hypertensive medications
  * Hospitalization for major cardiovascular- or hemodynamic-related events (such as heart failure or atrial fibrillation)
Incidence of serious adverse events (SAEs) related to the investigational device | From day 0 (procedure) to 12 months post index procedure
  The incident of serious adverse events (SAEs) related to the investigational device within 12 months post index procedure.
Incidence of device deficiency | At Visit 3, day 0 (procedure)
  Incidence of device deficiency
Mean ambulatory BP | From baseline at Visit 2 to 3- and 12-month post index procedure
  Changes from baseline in mean ambulatory BP including 24-hour ambulatory blood pressure, including ASBP and Ambulatory Diastolic Blood Pressure (ADBP), daytime and nighttime Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) measured by ABPM at 3- and 12-month post index procedure (except 24-hour mean daytime ASBP at 3-month post index procedure, which is already included in the primary endpoint)
Office blood pressure (OBP) | From baseline at Visit 2 to 1-, 3-, 6- and 12-month post index procedure
  Changes from baseline in office blood pressure (OBP) at 1-, 3-, 6- and 12-month post index procedure
Percentage of patients with office systolic blood pressure within target range | At 3-, 6- and 12-month post index procedure
  Percentage of patients with office systolic blood pressure (OSBP) within target range (SBP <140 mmHg and SBP <130 mmHg) at 3-, 6- and 12-month post index procedure
Percentage of patients with mean ASBP within the target range | At 3- and 12-month post index procedure
  Percentage of patients with mean ASBP within the target range (ASBP <130 mmHg) at 3- and 12-month post index procedure
Proportion of OSBP decreased by ≥ 5, 10, 15 and 20 mmHg | At 3-month post index procedure
  • The proportion of OSBP decreased by ≥ 5, 10, 15 and 20 mmHg at 3-month post index procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Barcelona Clinic Hospital, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Gao F, Ren C, Ma G, Bu P, Fu G, Chen H, Han Z, Li Y, Li J, Ma X, Hao L, Chen Y, Chen M, Chen X, Liu X, Jiang J, Yu J, Li N, Ma X, Yang B, Cong H, Wang X, Fan Q, Lv S, Wu D, Dai Q, Qiu F, Cai H, Zhou YJ. The Netrod six-electrode radiofrequency renal denervation system for uncontrolled hypertension: a sham-controlled trial. Eur Heart J. 2024 Nov 21;45(44):4761-4764. doi: 10.1093/eurheartj/ehae703. No abstract available. PMID 39431289